CLINICAL TRIAL: NCT00763971
Title: A Phase III, Randomised, Double-Blind, Multicentre, Parallel-Group, Placebo- and Active-Controlled, Dose-Optimisation Safety and Efficacy Study of Lisdexamfetamine Dimesylate (LDX) in Children and Adolescents Aged 6-17 With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Randomized, Double-blind Safety and Efficacy Study of Lisdexamfetamine Dimesylate (LDX) in Children and Adolescents Aged 6-17
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD489-325; 2008-000679-90 (EudraCT Number)
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Results first posted 2012-03-22 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate; Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Lisdexamfetamine Dimesylate (LDX) (Experimental): Overencapsulated LDX 30, 50, or 70mg
  Interventions: Drug: Lisdexamfetamine Dimesylate (LDX)
- Methylphenidate Hydrochloride (Active Comparator): Overencapsulated Concerta 18, 36, or 54mg
  Interventions: Drug: Methylphenidate Hydrochloride
- Placebo (Placebo Comparator): Overencapsulated Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lisdexamfetamine Dimesylate (LDX) — 30, 50 or 70mg capsule once per day (Overencapsulated)
  Other Names: Vyvanse™
  Arms: Lisdexamfetamine Dimesylate (LDX)
Drug: Methylphenidate Hydrochloride — 18, 36, or 54mg tablet one per day (Overencapsulated)
  Other Names: Concerta®, OROS MPH
  Arms: Methylphenidate Hydrochloride
Drug: Placebo — Placebo capsule once per day (Overencapsulated)
  Arms: Placebo

SUMMARY:
The main aim of this study is to see if giving LDX to children and adolescents aged 6-17 years with ADHD decreases symptoms of ADHD.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or female aged 6-17 years inclusive at the time of consent.
2. Subject must meet Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition - Text Revision (DSM-IV-TR) criteria for a primary diagnosis of ADHD based on a detailed psychiatric evaluation.
3. Subject must have a Baseline ADHD-RS-IV total score ≥28.
4. Subject has blood pressure measurements within the 95th percentile for age, gender, and height at Screening and Baseline.
5. Subject is able to swallow a capsule.

Exclusion Criteria:

1. Subject has failed to respond to more than one adequate course (dose and duration) of stimulant therapy. One course must have been a long-acting formulation.
2. Subject has a conduct disorder. Oppositional Defiant Disorder is not exclusionary.
3. Subject is currently considered a suicide risk, has previously made a suicide attempt or has a prior history of, or is currently, demonstrating active suicidal ideation.
4. Subject has glaucoma.
5. Subject weighs less than 22.7kg (50lbs).
6. Subject is significantly overweight based on Centre for Disease Control and Prevention Body Mass Index (BMI)-for-age gender specific charts at Screening. Significantly overweight is defined as a BMI >97th percentile for this study.
7. Subject has a documented allergy, hypersensitivity, or intolerance to amphetamine or methylphenidate.
8. Subject has a documented allergy, hypersensitivity, or intolerance to any excipients in the test or reference products.
9. Subject has a history of seizures (other than infantile febrile seizures), a tic disorder, or a current diagnosis and/or a known family history of Tourette's Disorder.
10. Subject has a known history of symptomatic cardiovascular disease, advance arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, or other serious cardiac problems that may place them at increased vulnerability to the sympathomimetic effects of a stimulant drug.
11. Subject has a known family history of sudden cardiac death or ventricular arrhythmia.
12. Subject is well controlled on their current ADHD medication with acceptable tolerability.
13. Subject has a pre-existing severe gastrointestinal tract narrowing (pathologic or iatrogenic).

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 336 (Actual)
Dates: Start 2008-11-17 (Actual); Primary Completion 2011-03-16 (Actual); Study Completion 2011-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (49):
- Belgium (3):
  - ZiekenhuisNetwerk Antwerpen, Commandant Weynsstraat 165, Campus Hoge Beuken, Hoboken, Antwerp
  - Universitair Ziekenhuis Gent, Kinder-en Jeugdpsychiatrie, De Pintelaan 185, Ghent, East Flanders
  - Afdeling Psychiatrie, UZ Herestraat 49, Bus 07003, Leuven
- France (4):
  - Hospital Archet 2, Nice, Cedex 03
  - Centre Hospitalier Charles Perrens, Bordeaux, Service de Psychiatrie de l'Enfant et de l'Adolescent, Bordeaux Cédex
  - Hôpital Gui de Chauliac, 80, avenue Augustin Fliche, Montpellier
  - Hôpital Robert Debré, Service de Psychopathologie de l'Enfant et de l'Adolescent, Paris, Île-de-France Region
- Germany (13):
  - Zentralinstitut für Seelische Gesundheit Mannheim, Klinik für Psychiatrie und Psychotherapie des Kindes-und Jug, J4/J5, Mannheim, Baden Wuttemburg
  - Schwerpunktpraxis für Entwicklung und Lernen, Heinrichsdamm 6, Bamberg, Bavaria
  - Medizinisches Studienzentrum Würzburg, Augustinerstrasse 10, Würzburg, Bavaria
  - Universität Würzburg, Klinik und Poliklinik fuer Kinder-und Jugendpsychiatrie und Psychotherapie, Würzburg, Bavaria
  - Universitatsklinikum Gießen und Marburg GmbH, Hans-Sachs-Strasse 4, Marburg, Hesse
  - Universitat Gottingen, Göttingen, Lower Saxony
  - Klinikum der Johannes Gutenberg-Universität Mainz, Klinik und Poliklinik für Kinder-und Jugendpsychiatrie und-psychotherapie,, Mainz, Rhineland-Palatinate
  - Universitätsmedizin Berlin, Berlin
  - Albert-Ludwigs-Universitat Freiburg, Freiburg im Breisgau
  - Praxis Dr. Walter Robert Otto, Fulda
  - Praxis Dr. Wolff, Hagen
  - Praxis Dr. med. Friedrich Kaiser und Dr. med. Ingrid Marinesse, Hamburg
  - Praxis für Neuropädiatrie, Schomburgstrasse 120, Hamburg
- Hungary (4):
  - Vadaskert Kórház és Szakambulancia, Budapest
  - Pándy Kálmán Kórház, Gyula
  - Gyermek és Ifjúságpszichiátriai Szakrendelés és Gondozó, Pécs
  - Szegedi Tudományegyetem, Szeged
- Italy (3):
  - Università degli Studi di Cagliari, Dipartimento di Neuroscienze, Cagliari
  - Azienda Ospedaliera Universitaria Policlinico G. Martino, Messina
  - Azienda Ospedaliera della 2 Universita di Napoli, Napoli
- Netherlands (2):
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Universitair Medisch Centrum Sint Radboud, Reinier Postlaan 10, Nijmegen
- Poland (4):
  - Szpital Uniwersytecki im. dr. Antoniego Jurasza w Bydgoszczy, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Wojewodzki Osrodek Lecznictwa Psychiatrycznego, Torun, Kuyavian-Pomeranian Voivodeship
  - Samodzielny Publiczny Dzieciecy Szpital Kliniczny, Warsaw, Masovian Voivodeship
  - Gdanski Uniwersytet Medyczna w Gdansku, Gdansk, Pomeranian Voivodeship
- Spain (7):
  - Hospital Sant Joan de Dèu, Esplugues de Llobregat, Barcelona
  - Hospital Marítimo, Unidad de Salud Mental Infanto-Juvenil (USMI-J), Carretera del Sanatorio s/n, Torremolinos, Malaga
  - Clínica Universitaria de Navarra, Unidad de Psiquiatría Infantil y Adolescente, Dept. de Psiquiatría y Psicología Médica, Pamplona, Navarre
  - Hospital Universitario de Canarias C/Ofra, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Complejo Hospitalario Universitario de Badajoz, Badajoz
  - Mutua de Terrassa, Barcelona
  - Hospital Ramón y Cajal, Servicio de psiquiatría, Madrid
- Sweden (4):
  - Utvecklingsneurologiska Enheten (UNE), BUC, Lockerudsv 12, Mariestad, Vastergotland
  - Drottning Silvias Barnsjukhus, Gothenburg
  - Astrid Lindgren Children's Hospital, Karolinska University Hospital, Stockholm
  - Barn och Ungdomsmedicin klinik Mölnlycke, Ekdalavägen 2,Box 9, Stockholm
- United Kingdom (5):
  - Basildon Hospital, Child Developement Centre, Nethermayne, Basildon, Essex
  - Lighthouse Child Development Centre, Snakes Lane, Southend-on-Sea, Essex
  - Victoria Hospital, Paediatric Unit, Hayfield Road, Kirkcaldy, Fife, Scotland
  - Tayside Childrens Hospital, Clinical Research Facility, Level 4, Dundee, Scotland
  - Ryegate Children's Centre, Tapton Crescent Road, Sheffield, Yorkshire

REFERENCES:
- [Result] Coghill D, Banaschewski T, Lecendreux M, Soutullo C, Johnson M, Zuddas A, Anderson C, Civil R, Higgins N, Lyne A, Squires L. European, randomized, phase 3 study of lisdexamfetamine dimesylate in children and adolescents with attention-deficit/hyperactivity disorder. Eur Neuropsychopharmacol. 2013 Oct;23(10):1208-18. doi: 10.1016/j.euroneuro.2012.11.012. Epub 2013 Jan 15. PMID 23332456
- [Result] Coghill DR, Banaschewski T, Lecendreux M, Zuddas A, Dittmann RW, Otero IH, Civil R, Bloomfield R, Squires LA. Efficacy of lisdexamfetamine dimesylate throughout the day in children and adolescents with attention-deficit/hyperactivity disorder: results from a randomized, controlled trial. Eur Child Adolesc Psychiatry. 2014 Feb;23(2):61-8. doi: 10.1007/s00787-013-0421-y. Epub 2013 May 25. PMID 23708466
- [Result] Banaschewski T, Soutullo C, Lecendreux M, Johnson M, Zuddas A, Hodgkins P, Adeyi B, Squires LA, Coghill D. Health-related quality of life and functional outcomes from a randomized, controlled study of lisdexamfetamine dimesylate in children and adolescents with attention deficit hyperactivity disorder. CNS Drugs. 2013 Oct;27(10):829-40. doi: 10.1007/s40263-013-0095-5. PMID 23893527
- [Derived] Setyawan J, Yang H, Cheng D, Cai X, Signorovitch J, Xie J, Erder MH. Developing a Risk Score to Guide Individualized Treatment Selection in Attention Deficit/Hyperactivity Disorder. Value Health. 2015 Sep;18(6):824-31. doi: 10.1016/j.jval.2015.06.005. Epub 2015 Aug 20. PMID 26409610
- See also: FDA recal information — http://www.fda.gov/opacom/7alerts.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Lisdexamfetamine Dimesylate (LDX): Lisdexamfetamine Dimesylate (LDX, Vyvanse®, SPD489) was administered orally once-daily at approximately 7:00AM for 7 weeks (4-week dose optimization period and a 3-week dose maintenance period) at doses of either 30, 50, or 70 mg.
- Methylphenidate Hydrochloride: Methylphenidate Hydrochloride (Concerta®, OROS MPH) was administered orally once-daily at approximately 7:00AM for 7 weeks (4-week dose optimization period and a 3-week dose maintenance period) at doses of either 18, 36, or 54 mg.
- Placebo: Placebo was administered orally once-daily at approximately 7:00AM for 7 weeks.
Period: Overall Study
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Methylphenidate Hydrochloride | Placebo
Started | 113 | 112 | 111
Completed | 80 | 74 | 42
Not Completed | 33 | 38 | 69
Not completed — Adverse Event | 5 | 2 | 4
Not completed — Protocol Violation | 3 | 3 | 2
Not completed — Withdrawal by Subject | 4 | 5 | 5
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Lack of Efficacy | 11 | 22 | 54
Not completed — Unable to swallow capsule | 2 | 1 | 1
Not completed — Personal reason | 3 | 0 | 0
Not completed — Exclusion criteria met | 1 | 0 | 0
Not completed — Sponsor decision | 1 | 0 | 0
Not completed — Due to holiday season | 2 | 0 | 1
Not completed — Randomization error | 0 | 0 | 1
Not completed — Medical monitor decision | 0 | 0 | 1
Not completed — Moved to another country | 0 | 1 | 0
Not completed — Subject wanted dose reduction | 0 | 1 | 0
Not completed — Lack of availability | 0 | 1 | 0
Not completed — Performed final visit on phone | 0 | 1 | 0
Not completed — Participation in 489-326 required | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Methylphenidate Hydrochloride | Placebo | Total
Number analyzed (Participants) | 111 | 111 | 110 | 332
Age, Continuous [Mean (Standard Deviation); unit: years] — Safety Population was used for demographics. Safety Population defined as all subjects who took at least 1 dose of investigational product. Four randomized subjects (2 in the LDX group, 1 in the Methylphenidate group, and 1 in the placebo group) did not receive investigational product and were therefore excluded from the Safety Population (n = 332).
  years | 10.9 (2.87) | 10.9 (2.63) | 11.0 (2.82) | 10.9 (2.77)
Age, Customized [Count of Participants; unit: Participants] — Safety Population was used for demographics. Safety Population defined as all subjects who took at least 1 dose of investigational product. Four randomized subjects (2 in the LDX group, 1 in the Methylphenidate group, and 1 in the placebo group) did not receive investigational product and were therefore excluded from the Safety Population (n = 332).
  Participants
    6-12 years | 77 | 80 | 79 | 236
    13-17 years | 34 | 31 | 31 | 96
Sex: Female, Male [Count of Participants; unit: Participants] — Safety Population was used for demographics. Safety Population defined as all subjects who took at least 1 dose of investigational product. Four randomized subjects (2 in the LDX group, 1 in the Methylphenidate group, and 1 in the placebo group) did not receive investigational product and were therefore excluded from the Safety Population( n = 332).
  Participants
    Female | 24 | 21 | 19 | 64
    Male | 87 | 90 | 91 | 268
Region of Enrollment [Count of Participants; unit: Participants] — This includes All Enrolled Subjects. Enrolled Population defined as all subjects who were randomized (n = 336).
  Participants
    France | 10 | 9 | 11 | 30
    Hungary | 11 | 10 | 11 | 32
    Spain | 13 | 14 | 14 | 41
    Poland | 3 | 4 | 3 | 10
    Belgium | 4 | 3 | 4 | 11
    Netherlands | 1 | 0 | 0 | 1
    Germany | 36 | 36 | 35 | 107
    United Kingdom | 8 | 10 | 9 | 27
    Italy | 9 | 9 | 7 | 25
    Sweden | 18 | 17 | 17 | 52

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Attention Deficit Hyperactivity Disorder Rating Scale-fourth Edition (ADHD-RS-IV) Total Score at up to 7 Weeks
Description: The ADHD-RS-IV consists of 18 items scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms) with total score ranging from 0 to 54. A decrease in score indicates an improvement in ADHD symptomology.
Time Frame: Baseline and up to 7 weeks
Population: Full Analysis set (FAS) defined as all subjects who were randomized and who took at least 1 dose of investigational product.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Methylphenidate Hydrochloride | Placebo
Number analyzed (Participants) | 98 | 103 | 104
Scores on a scale | -24.3 (1.16) | -18.7 (1.14) | -5.7 (1.13)
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate (LDX) vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; difference in LS means = -18.6, 95% CI 2-sided [-21.5 to -15.7]
Statistical Analysis 2: Comparison: Methylphenidate Hydrochloride vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; difference in LS means = -13.0, 95% CI 2-sided [-15.9 to -10.2]

2. Secondary Outcome: Percentage of Participants With Improvement on Clinical Global Impression-Improvement (CGI-I) Scores
Description: Clinical Global Impression-Improvement (CGI-I) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: Up to 7 weeks
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Methylphenidate Hydrochloride | Placebo
Number analyzed (Participants) | 100 | 104 | 104
percentage of participants | 78.0 | 60.6 | 14.4
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate (LDX) vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; difference in percentages = 63.6, 95% CI 2-sided [53.0 to 74.1]
Statistical Analysis 2: Comparison: Methylphenidate Hydrochloride vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; difference in percentages = 46.2, 95% CI 2-sided [34.6 to 57.7]

3. Secondary Outcome: Change From Baseline in Conner's Parent Rating Scale - Revised (CPRS-R) Total Score at up to 7 Weeks
Description: The Conner's Parent rating Scale-revised short version (CPRS-R) consists of 27 questions graded on a scale from 0 (not true at all) to 3 (very much true) with a total score ranging from 0 to 81. Higher scores are indicative of increased ADHD. This scale allows parents to respond on the basis of the child's behavior and help assess ADHD and evaluate problem behavior.
Time Frame: Baseline and up to 7 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Methylphenidate Hydrochloride | Placebo
Number analyzed (Participants) | 96 | 99 | 100
Scores on a scale | -24.5 (1.70) | -18.4 (1.69) | -3.2 (1.69)
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate (LDX) vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; difference in LS means = -21.3, 95% CI 2-sided [-25.5 to -17.0]
Statistical Analysis 2: Comparison: Methylphenidate Hydrochloride vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; difference in LS means = -15.1, 95% CI 2-sided [-19.3 to -10.9]

4. Secondary Outcome: Health Utilities Index-2 (HUI-2) Scores at up to 7 Weeks
Description: HUI is used to describe health status and to obtain utility scores by collecting data using one or more questionnaires in formats selected to match the specific study design criteria. Scoring ranges from 0.00 (dead) to 1.00 (perfect health). Higher scores represent better health status.
Time Frame: Baseline and up to 7 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Methylphenidate Hydrochloride | Placebo
Number analyzed (Participants) | 98 | 103 | 97
Scores on a scale
  Baseline | 0.811 (0.1451) | 0.822 (0.1377) | 0.806 (0.1460)
  Up to 7 weeks | 0.878 (0.1322) | 0.887 (0.1151) | 0.843 (0.1431)

5. Secondary Outcome: Change From Baseline in the Child Health and Illness Profile, Child Edition: Parent Report Form (CHIP-CE:PRF) Global T-score at up to 7 Weeks
Description: The CHIP-CE:PRF evaluates health-related quality of life. It is composed of 5 domains (satisfaction, comfort, resilience, avoidance, and achievement) consisting of a total of 76 items. The global score is an average of the scores for the 5 domains. The majority of items assess frequency of events using a 5-point response format. There is no range for a total score. Raw scale scores are used to generate T-scores. Higher scores indicate better health.
Time Frame: Baseline and up to 7 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: T-scores
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Methylphenidate Hydrochloride | Placebo
Number analyzed (Participants) | 78 | 75 | 80
T-scores | 8.6 (1.08) | 7.1 (1.10) | -0.2 (1.07)
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate (LDX) vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; difference in LS means = 8.8, 95% CI 2-sided [6.1 to 11.5]
Statistical Analysis 2: Comparison: Methylphenidate Hydrochloride vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; difference in LS means = 7.3, 95% CI 2-sided [4.6 to 10.0]

6. Secondary Outcome: Change From Baseline in Weiss Functional Impairment Rating Scale - Parent Report (WFIRS-P) Global Score at up to 7 Weeks
Description: The WFIRS-P is a 50-item scale with each item scored from 0 (never/not at all) to 3 (very often/very much). Mean scores range from 0 to 3. Higher scores indicate greater functional impairment.
Time Frame: Baseline and up to 7 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Methylphenidate Hydrochloride | Placebo
Number analyzed (Participants) | 79 | 83 | 87
Scores on a scale | -0.3 (0.04) | -0.3 (0.04) | 0.0 (0.04)
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate (LDX) vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; difference in LS means = -0.3, 95% CI 2-sided [-0.4 to -0.2]
Statistical Analysis 2: Comparison: Methylphenidate Hydrochloride vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; difference in LS means = -0.2, 95% CI 2-sided [-0.3 to -0.1]

7. Secondary Outcome: Change From Baseline in Brief Psychiatric Rating Scale for Children (BPRS-C) Total Score at up to 7 Weeks
Description: The BPRS-C characterizes psychopathology. A total of 21 items are rated on a scale from 0 (not present) to 6 (extremely severe) with a total score ranging from 0 to 126. A decrease in score indicates a reduction in psychopathology.
Time Frame: Baseline and up to 7 weeks
Population: Safety Population defined as all subjects who took at least 1 dose of investigational product.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Methylphenidate Hydrochloride | Placebo
Number analyzed (Participants) | 20 | 21 | 22
Scores on a scale | -9.15 (11.264) | -9.71 (6.936) | -2.59 (7.436)

8. Secondary Outcome: Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS is a 19-item semi-structured interview designed to capture suicide-related thoughts and behaviors.
Time Frame: Up to 7 weeks
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Methylphenidate Hydrochloride | Placebo
Number analyzed (Participants) | 25 | 29 | 27
participants
  Suicidal ideation | 1 | 0 | 0
  Non-suicidal self injurious behavior | 1 | 0 | 0

ADVERSE EVENTS:
Description: Safety Population defined as all subjects who took at least 1 dose of investigational product.
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Methylphenidate Hydrochloride | Placebo
Serious Adverse Events (participants affected / at risk) | 3/111 | 2/111 | 3/110
Other Adverse Events (participants affected / at risk) | 80/111 | 72/111 | 63/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lisdexamfetamine Dimesylate (LDX) (N=111) | Methylphenidate Hydrochloride (N=111) | Placebo (N=110)
Syncope (Nervous system disorders) | 1 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Loss of conciousness (Nervous system disorders) | 0 | 0 | 1
Hematoma (Vascular disorders) | 0 | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lisdexamfetamine Dimesylate (LDX) (N=111) | Methylphenidate Hydrochloride (N=111) | Placebo (N=110)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 4 (4) | 6 (10)
Abdominal upper pain (Gastrointestinal disorders) | 8 (15) | 9 (10) | 6 (9)
Diarrhea (Gastrointestinal disorders) | 5 (8) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 12 (14) | 8 (8) | 3 (4)
Vomiting (Gastrointestinal disorders) | 4 (5) | 4 (4) | 1 (1)
Fatigue (General disorders) | 5 (5) | 1 (1) | 3 (3)
Irritability (General disorders) | 4 (6) | 4 (5) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 5 (5) | 0 (0)
Gastroenteritis (Infections and infestations) | 4 (4) | 3 (3) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 8 (9) | 14 (14) | 8 (9)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1) | 2 (2)
Joint sprain (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) | 1 (1)
Wrong drug administered (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 3 (7) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 15 (15) | 5 (5) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 12 (13) | 6 (8) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 28 (31) | 17 (21) | 3 (3)
Dizziness (Nervous system disorders) | 4 (4) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 16 (21) | 22 (30) | 22 (27)
Migraine (Nervous system disorders) | 3 (4) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 4 (4) | 3 (3) | 1 (1)
Initial insomnia (Psychiatric disorders) | 3 (3) | 7 (7) | 1 (1)
Insomnia (Psychiatric disorders) | 16 (16) | 9 (9) | 0 (0)
Sleep disorder (Psychiatric disorders) | 6 (6) | 2 (2) | 1 (1)
Tic (Psychiatric disorders) | 2 (2) | 3 (4) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (8) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.